CLINICAL TRIAL: NCT04438785
Title: Effects of Myofunctional Therapy With an M-health Application Airway Gym in Severe Apnea/Hypopnea Sleep Obstructive Syndrome: A Randomized Multicentre Control Trial
Brief Title: Effects of Myofunctional Therapy With an Application in Severe Apnea/Hypopnea Sleep Obstructive Syndrome (MTASSAOS)
Acronym: MTASSAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quironsalud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90694424
Record Dates: First submitted 2020-06-09; First posted 2020-06-19 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-06

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: SEVERE OSAHS; MYOFUNTIONAL THERAPY; M HEALTH APPLICATION; TELEMEDICINE
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Interventional prospective multicentre trial with consecutive random assignment
Who Masked: Outcomes Assessor
Masking Description: Results will be analysed blinded by the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (AirwayGym) GROUP (Experimental): Patients newly diagnosed with severe OSAHS should perform muscle upper airway exercises using the AirwayGym app for 20 min a day for 90 days.
  Interventions: Device: The intervention consists of myofunctional therapy (MT) using the AirwayGym app.
- CONTROL GROUP (No Intervention): Patients newly diagnosed with severe OSAHS do no therapy for 90 days.

INTERVENTIONS:
Device: The intervention consists of myofunctional therapy (MT) using the AirwayGym app. — Intervention. Patient newly diagnosed with severe OSAHS should perform muscle upper airway exercises using the App AirwayGym 20 minutes a day during 90 days.
  Arms: INTERVENTION (AirwayGym) GROUP

SUMMARY:
• Background and study aims: Obstructive sleep apnea is a potentially serious sleep disorder. It causes breathing to stop and start repeatedly during sleep. There are several types of sleep apnea, the most common of which is obstructive sleep apnea. This type of apnea occurs when an individual's throat muscles intermittently relax and block the airway during sleep.

The classic treatment for this disease is based on weight loss, and exercise, and the use of a continuous positive airway pressure (CPAP) machine.

Myofunctional therapy (MT) is one of the newest treatments for sleep-disordered breathing. MT is based on daily exercises of the throat muscles in an attempt to strengthen them and facilitate opening of the airway.

Who can participate? Patients diagnosed with severe sleep apnea and aged between 18-75 years.

What does the study involve? Participants will be randomly allocated to either use of the "AirwayGym" smartphone app or no treatment for 3 months. The AirwayGym app provides instructions on how to perform exercises to strengthen the throat muscles and reminds participants to perform the exercises for 20 min per day. Participants will be assessed monthly at the clinic.

What are the possible benefits and risks of participating? Benefits: Curing sleep apnea syndrome. There are no significant risks for participants.

Where is the study run from? Hospital Quirónsalud Marbella (Spain) When is the study starting and how long is it expected to run for? October 2018 to January 2021 Who is funding the study? Investigator initiated and funded Who is the main contact? Dr. Carlos O'Connor Reina, coconnor@us.es

DETAILED DESCRIPTION:
INTRODUCTION Obstructive sleep apnea/hypopnea syndrome (OSAHS) has become one of the more serious health problems worldwide (Mendes et al., 2014). Because of its relationship with obesity, its prevalence and incidence have increased. It is associated with morbidities such as cardiovascular and cerebrovascular diseases. The classic treatment of this disease is based on dietary measures, weight loss, and exercise, and the use of a continuous positive airway pressure (CPAP) machine.

Myofunctional therapy (MT) is one of the newest treatments for sleep-disordered breathing (Camacho et al., 2015). MT is based on daily exercises using the oropharyngeal muscles in an attempt to strength them and facilitate opening of the airway. OSAHS originates from the suboptimal function of the dilator muscles of the airway. Therefore, MT is a therapy designed theoretically to deal with the underlying mechanism of this disease (Korhan et al., 2015). MT is based on oropharyngeal exercises described by diagrams, videos, and weekly instructions from a myofunctional therapist. The patient is instructed to perform the exercises regularly, for at least 3 months, and for 30 min daily. In some cases, patients perform exercises by themselves at home without substantial feedback and without giving precise information to the therapist about their performance of the exercises (O'Connor et al., 2019).

Most existing mobile health (mHealth) apps for OSAHS focus on diagnosis of snoring or OSAHS (Isetta et al., 2017), while a few are designed to promote adherence to treatment with CPAP (Camacho et al., 2015). To our knowledge, there are no apps that focus on the treatment of OSAHS. However, mobile technology could be especially valuable in treating OSAHS patients because of its potential to promote patient empowerment and self-management (Iftikhar et al., 2017).

One of the best treatments for OSAHS is exercise and weight loss (Iftikhar et al., 2018). Because patients' time is limited, the investigators consider that there will be a greater probability of their performing the exercises if they are able to do wherever and whatever. Therefore, the investigators designed and developed a novel mHealth app to promote oropharyngeal exercises while interacting with a smartphone. In this prospective randomized multicenter clinical trial, the investigators aim to evaluate adherence to the app and its effectiveness in a group of patients (AirwayGym group, AGG) with severe OSAHS compared with a control group (CG) of similar patients.

HYPOTHESIS The regular use of the AirwayGym app, which is designed to perform and increase adherence to MT, will improve OSAHS in patients with severe disease ,apnea hypopnea index (AHI)>30) by increasing the tone of their upper airway muscles.

OBJECTIVES The main objective will be to study the evolution of the use of the app based on MT in patients diagnosed with severe OSAHS.

Secondary Objectives:

1. To evaluate the influence of MT using an app on the change in the AHI in patients diagnosed with severe OSAHS.
2. To evaluate O2 nadir and O2 desaturation index.
3. To use scores obtained using the Iowa Oral Performance Instrument (IOPI) to evaluate the tone of genioglossus and buccinator muscles.
4. To evaluate subjective morning somnolence and sleep quality score using the Epworth Sleepiness Scale and Pittsburgh Sleep Quality Index.

METHODS Design: Prospective controlled quasi-experimental clinical trial in patients with severe OSAHS (AHI>30). Study population: Patients recently diagnosed with severe OSAHS who agree to participate in this clinical trial.

Evaluation of the effectiveness of use of the app in performing MT in patients with severe OSAHS will be performed using the longitudinal values obtained during study, based on the percentage of improvement in the AHI observed during follow-up. This percentage has been calculated from results reported in previous MT studies published and presented in the bibliography. To achieve a confidence level of 95% and power of 80% with an estimated improvement of the AHI of 60%, the required sample size is 30 patients (15 AirwayGym group [AGG], 15 CG).

Randomization will be based on the consecutive order of patient enrollment, with odd numbers allocated to the AGG (patients treated with the app) and even numbers to the CG (patients without complementary therapy).

Patients without a smartphone will be directly recruited to the CG. VARIABLES EVALUATED: Age, sex, weight, height, body mass index (BMI), waist circumference (belly button height), neck circumference, IOPI lingual and buccinator, AHI, O2 desaturation index, and O2 nadir.

Questionnaires: Friedman stage, Epworth Sleepiness Scale, and Pittsburgh Sleep Quality Index PROCEDURE The AGG will use the app, which was created in a collaboration between the Sleep Units of Hospital Quirónsalud Marbella and Campo de Gibraltar. The novelty of this app is that it is the first in the healthcare market in which the patient can interact directly with the smartphone; the phone provides acoustic feedback about the efficacy of the exercises performed and is focused on sleep apnea disease and improving proprioceptive deficits. The app includes nine exercises based on MT that attempt to enhance the tonicity of the various muscles involved in the pathogenesis of OSAHS. Before every exercise, an animated demonstration and a video show the patient how to perform the exercise. At the conclusion of each exercise, the patient receives feedback about the success of their performance via a point score. When the patient finishes the exercises, they are saved in the cloud and a therapist can evaluate the performance of them. A chat function is available where patient can contact the therapist.

This app complies with regulation 2002/58/Community European (CE) and (UE) 2016/679 concerning data protection.

The main objective of these exercises is to increase the tone of the extrinsic muscles of the tongue.

The exercises are based on those described elsewhere (Guimaraes et al., 2009), adapted to obtain feedback with the phone and to stimulate proprioceptive sensors with acoustic feedback.

For hygiene reasons, it is recommended that participants cover the screen with cling film during all exercises.

The CG does not use any therapy for OSAHS for 3 months. All patients will attend hospital once a month for measurement of the variables (weight, height, BMI, neck and waist circumference, completion of the questionnaires, IOPI scores)

Schedule of visits:

SELECTION VISIT Patients with newly diagnosed severe OSAHS based on home or laboratory polygraphy with measures of AHI, O2 saturation, and O2 nadir were evaluated. All sleep studies were manually interpreted by a sleep technician according to the standard criteria of the American Academy of Sleep Medicine (AASM) Manual for the Scoring of Sleep and Associated Events, and were reviewed by certified physicians. Information about inclusion and exclusion criteria, evaluation of the type of smartphone used, previous experience with the app, and the study protocol was provided. After any questions were resolved, the patient agreed to participate and signed informed consent (IC).

INITIAL VISIT Participants were evaluated by an Ear nose and throat (ENT) specialist and underwent pharyngoscopy, rhinofibrolaryngoscopy, Friedman staging, Marchesani protocol, and examination of their temporomandibular joint dysfunction. If the patient presented with tonsillitis grade IV, complete nose obstruction, ankyloglossia, or problems with temporomandibular joint dysfunction, they were excluded from the study.

SECOND VISIT: Variables were measured (weight, height, BMI, neck and waist circumference, completion of questionnaires, IOPI scores) and randomization was performed to AGG or CG. Participants in the AGG were instructed about the use of the app and the exercises to do.

FOLLOW-UP VISITS:

AGG: Participants performed exercises daily for about 20 min. Follow-up visits occurred after 1 month (visit 3) and 3 months (visit 4). At these visits, variables were measured, questionnaires completed, and exercise performance checked.

CG: Follow-up visits occurred after 1 month (visit 3) and 3 months (visit 4). At these visits, variables were measured, questionnaires completed, and it was checked that no other therapies are being followed.

Final visit: At 3 months for both groups. At this visit, questionnaires were completed, variables were measured again, and laboratory or in-home polygraphy was performed. The total study duration for each participant was 3 months.

DISCONTINUATION CRITERIA

A participant in either group was excluded from the study if:

1. They did not perform exercises during at least 85% of the scheduled sessions,or were lost to follow-up because they did not attend hospital visits.
2. They lost 5% of their body weight during study participation. Data were collected in a database. Nominal variables were described by their frequency distribution. Quantitative variables were assessed by calculating the arithmetic mean and standard deviation. Baseline characteristics of the two groups of participants with OSAHS were compared by two-tailed paired t tests for continuous variables and chi-squared or Fisher's exact test for nominal variables. For variables with skewed distribution, the investigators performed Mann-Whitney tests. In addition, the investigators performed Pearson correlation analysis of changes in AHI compared with changes in possible explanatory variables, including BMI and neck and waist circumference. A P value less than 0.05 was considered significant.

The main outcome measures are polygraphy findings at the beginning and end of the study, IOPI scores at the beginning and end of the study, Epworth Sleepiness Scale and Pittsburgh Sleep Quality Index at all visits, weight in kg, height in cm, BMI in kg/m2, and neck and waist circumference in cm at all visits.

ETHICAL APPROVAL After evaluating and revising the protocol, the Investigation Ethical Committee (EC) from Costa del Sol approved the study with the code AWGAPN-2019-01. Before starting the trial, all participants had to have signed and dated all IC approved by the EC.

Access to data and data protection. To ensure confidentiality of study data, the original data were stored in the Hospital and only the investigators and the Investigation EC had access.

UTILITY This app could improve participants' AHI and quality of life and reduce their clinical symptoms and need for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Recently diagnosed with severe sleep apnea and do not have any previous experience or information with this pathology
* Consent signed

Exclusion Criteria:

* BMI > 40 kg/m²
* Inability to fill up questionnaires
* Severe drug or alcohol abuse
* Hypnotic medication
* Not controlled coronary disease
* Decompensated Heart failure
* Stroke
* Systemic Disease associated with inflammatory diagnosed entity (arthritis, sarcoidosis, vasculitis, lupus…)
* Neuromuscular disease (like Duchenne)
* Craniofacial deformities.
* Active oncologic process.
* Any antecedents of MT treatment or other treatment for sleep apnea could affect study results of the study (surgery, Mandibular Advancement Device (MAD) or CPAP).

Once the patient accepted and signed consent and met inclusion criteria, they will be attended by Ent specialist to rule out:

* Severe upper airway obstruction (Complete nose obstruction, Tonsils grade IV/IV )
* Presence of tongue tie (Marchesani protocol) with limitation of tongue movements
* Antecedents or presence of temporomandibular joint disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JOSE MARIA IGNACIO GARCIA, MD, Study Chair — NEUMOLOGY DEPARMENT HOSPITAL QUIRONSALUD MARBELLA; FRANCISCO JESUS GONZALEZ SANCHEZPharm D, Pharm D, Study Director — RESEARCH UNIT HOSPITAL QUIRONSALUD MARBELLA; CARLOS O´CONNOR REINA, MD, Principal Investigator — OTOLARINGOLOGY DEPARMENT HOSPITAL QUIRONSALUD MARBELLA
Locations (2):
- Spain (2):
  - Hospital Quironsalud Campo de Gibraltar, Los Barrios, Cadiz
  - Hospital Quironsalud Marbella, Marbella, Malaga

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not expected to be made available due to confidentiality

REFERENCES:
- [Background] Mendes FA, Marone SA, Duarte BB, Arenas AC. Epidemiologic profile of patients with snoring and obstructive sleep apnea in a university hospital. Int Arch Otorhinolaryngol. 2014 Apr;18(2):142-5. doi: 10.1055/s-0033-1359309. Epub 2014 Feb 28. PMID 25992080
- [Background] Camacho M, Certal V, Abdullatif J, Zaghi S, Ruoff CM, Capasso R, Kushida CA. Myofunctional Therapy to Treat Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. Sleep. 2015 May 1;38(5):669-75. doi: 10.5665/sleep.4652. PMID 25348130
- [Background] Korhan I, Gode S, Midilli R, Basoglu OK. The influence of the lateral pharyngeal wall anatomy on snoring and sleep apnoea. J Pak Med Assoc. 2015 Feb;65(2):125-30. PMID 25842544
- [Background] Isetta V, Torres M, Gonzalez K, Ruiz C, Dalmases M, Embid C, Navajas D, Farre R, Montserrat JM. A New mHealth application to support treatment of sleep apnoea patients. J Telemed Telecare. 2017 Jan;23(1):14-18. doi: 10.1177/1357633X15621848. Epub 2016 Jul 8. PMID 26672606
- [Background] Camacho M, Robertson M, Abdullatif J, Certal V, Kram YA, Ruoff CM, Brietzke SE, Capasso R. Smartphone apps for snoring. J Laryngol Otol. 2015 Oct;129(10):974-9. doi: 10.1017/S0022215115001978. Epub 2015 Sep 3. PMID 26333720
- [Background] Iftikhar IH, Bittencourt L, Youngstedt SD, Ayas N, Cistulli P, Schwab R, Durkin MW, Magalang UJ. Comparative efficacy of CPAP, MADs, exercise-training, and dietary weight loss for sleep apnea: a network meta-analysis. Sleep Med. 2017 Feb;30:7-14. doi: 10.1016/j.sleep.2016.06.001. Epub 2016 Jun 28. PMID 28215266
- [Background] Iftikhar IH, Roland J. Obesity Hypoventilation Syndrome. Clin Chest Med. 2018 Jun;39(2):427-436. doi: 10.1016/j.ccm.2018.01.006. PMID 29779600
- [Result] O'Connor Reina C, Plaza Mayor G, Ignacio-Garcia JM, Baptista Jardin P, Garcia-Iriarte MT, Casado-Morente JC. Floppy Closing Door Epiglottis Treated Successfully with an Mhealth Application Based on Myofunctional Therapy: A Case Report. Case Rep Otolaryngol. 2019 Jul 1;2019:4157898. doi: 10.1155/2019/4157898. eCollection 2019. PMID 31355035
- [Result] O'Connor-Reina C, Ignacio Garcia JM, Rodriguez Ruiz E, Morillo Dominguez MDC, Ignacio Barrios V, Baptista Jardin P, Casado Morente JC, Garcia Iriarte MT, Plaza G. Myofunctional Therapy App for Severe Apnea-Hypopnea Sleep Obstructive Syndrome: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 9;8(11):e23123. doi: 10.2196/23123. PMID 33093013

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Started | 20 | 20
Completed | 18 | 10
Not Completed | 2 | 10
Not completed — change of weight, give up intervention | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.17 [56.4 to 71.3] | 63.9 [53.7 to 64.6] | 62.2 [54.5 to 68.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 14 | 8 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
IOPI tongue strength (is the maximun strength obtained by contraction of genioglossus muscle) [Median (Inter-Quartile Range); unit: kilopascals] | 39.83 [35.32 to 45.2] | 42 [32.6 to 51.3] | 41.3 [33.3 to 49.3]
IOPI Lip Strength (maximal lip strength measured with muscle buccinator) [Median (Inter-Quartile Range); unit: kilopascals] | 27.8 [24.1 to 32.4] | 28.1 [23.7 to 32.5] | 27.95 [23.9 to 32.4]

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: Measurement of number of apneas or hypopneas recorded during the study per hour of sleep
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
events per hour
  Apnea Hypopnea Index (BASELINE) | 44.77 [33.84 to 55.69] | 47.36 [38.59 to 56.13]
  Apnea Hypopnea Index(AFTER 3 MONTHS) | 20.88 [14.02 to 27.74] | 35 [31.2 to 38.7]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the Apnea Hypopnea Index from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 2.58

2. Primary Outcome: Evaluation of O2 Desaturation Index (ODI)
Description: The ODI is the number of times per hour of sleep that the blood oxygen level drops by a certain degree from baseline. Any respiratory event during sleep with a 3% drop in blood oxygen levels is counted towards the total. For example, a change from 95% to 92% would be an event that is counted toward the index's total.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
events per hour
  ODI (BASELINE) | 36.31 [27.19 to 43.43] | 40.64 [29.46 to 51.81]
  ODI (AFTER 3 MONTHS | 19.4 [12.9 to 25.98] | 32.03 [24.14 to 39.91]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the O2 desaturation index (ODI) from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.003, t-test, 2 sided; Median Difference (Final Values) = -0.971

3. Secondary Outcome: Evaluation of Iowa Oral Performance Instrument (IOPI) Score
Description: The IOPI objectively measures maximum tongue strength in kilopascals and represents the tone of the genioglossus muscles.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: Kilopascals
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
Kilopascals | 44.1 [39.5 to 48.8] | 31.3 [26.6 to 35.9]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the IOPI tongue score from baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Net) = -0.364

4. Secondary Outcome: Iowa Oral Performance Instrument Lip Strength
Description: The IOPI objectively measures maximum lip strength in kilopascals and represents the tone of the buccinator muscles.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: kilopascals
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
kilopascals
  IOPI Lip BASELINE | 27.89 [24.16 to 32.47] | 28.1 [23.7 to 32.5]
  IOPI Lip AFTER 3 MONTHS | 44.11 [39.5 to 48.8] | 31.3 [26.6 to 35.9]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the IOPI lip score from the baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.001, t-test, 2 sided; Median Difference (Final Values) = -1.131

5. Secondary Outcome: Neck Circumference (cm)
Description: Gives an idea if there is an anatomical change or reduction in fat in the upper airway muscles after intervention .
Time Frame: Baseline and three months.
Measure: Median (Inter-Quartile Range); unit: centimetres
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
centimetres
  Neck Circumference BASE LINE (CM) | 43.7 [41.03 to 46.4] | 43.7 [40.33 to 46.6]
  Neck Circumference 3 MONTHS (CM) | 44.6 [42.12 to 47.2] | 43.5 [40.33 to 46.67]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the neck circumference from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = 0.98

6. Secondary Outcome: Waist Circumference (cm)
Description: Gives an idea if there is an anatomical change or reduction of fat in the thorax muscles after intervention.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: centimetres
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
centimetres
  Waist circumference baseline (cm) | 109.2 [102.9 to 115.4] | 109.1 [97.5 to 120.6]
  Waist circumference after 3 months (cm) | 108.84 [102.9 to 115.4] | 108.5 [96.9 to 120.1]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the waist circumference from baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = 0.98

7. Secondary Outcome: Body Mass Index BMI
Description: is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass in kilograms divided by the square of the body height in meters, and is expressed in units kg/m^2 .
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: kilograms/m^2
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
kilograms/m^2
  BMI BASELINE kg/m^2 . | 28.9 [26.8 to 31.02] | 29.6 [27.1 to 32.08]
  BMI AFTER 3 MONTHS kg/m^2 . | 28.8 [26.7 to 30.8] | 29.6 [27.3 to 31.8]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP vs CONTROL GROUP; Evaluate if the BMI from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.97

8. Secondary Outcome: Epworth Sleepiness Scale
Description: A scale (0-24), obtained by self-administered questionnaire, that rates an individual's probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that people experience in their daily lives.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
score on a scale
  Epworth sleepiness scales (Baseline) | 10.3 [8.71 to 12.24] | 9.3 [6.6 to 12.11]
  Epworth sleepiness scales (Three months) | 5.3 [3.45 to 7.2] | 9.6 [6.8 to 12.3]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the Epworth Sleepiness Scale from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.001, t-test, 2 sided; Median Difference (Final Values) = -1.23

9. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: A scale (0- 21) obtained by a self-report questionnaire that assesses sleep quality over a 1-month time interval. The questionnaire consists of a combination of Likerttype and open-ended questions (later converted to scaled scores using provided guidelines).
  Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.A global score of 5 or more indicates poor sleep quality and that the higher the score, the worse the quality of sleep. The questionnaire consists of 19 individual items, creating seven components that produce one global score, and takes 5-10 min to complete.
Time Frame: Baseline and three months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
Number analyzed (Participants) | 18 | 10
score on a scale
  Pittsburgh sleep quality index (Baseline) | 10.2 [8.22 to 12.0] | 8.8 [7.1 to 10.48]
  Pittsburgh sleep quality index (Three Months) | 10.3 [8.71 to 12.2] | 9.78 [7.2 to 12.1]
Statistical Analysis 1: Comparison: INTERVENTION (AirwayGym) GROUP; Evaluate if the Pittsburgh sleep quality index from Baseline and after three months in the Intervention Group showed statistical significant difference p<0.05; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.98

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the performance of the study 3 months
Description: The definition of adverse event did not differ from Adverse Event definition. Event collection was done through daily telemedicine approach.
Arm/Group | INTERVENTION (AirwayGym) GROUP | CONTROL GROUP
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/10
Other Adverse Events (participants affected / at risk) | 0/18 | 0/10

LIMITATIONS AND CAVEATS:
In the end, we had a small sample recruited mainly due to Covid restrictions. We have a significant loss of patients in the control group (50%) due the severity of the disease and the need of therapy. Initially we start to perform polysomnographies but we change to polygraphies due to hospital needs during pandemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04438785/Prot_SAP_000.pdf